CLINICAL TRIAL: NCT00694863
Title: Treatment With Synthetic Adrenocorticotropic Hormone (ACTH) in Patients With Membranous Nephropathy and High Risk for Renal Failure. A Pilot Study
Brief Title: Treatment With Synthetic ACTH in High Risk Patients With Membranous Nephropathy
Acronym: ACTHiMeN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008.1; ABR: NL22482.091.08; CMO: 2008/77
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2010-12

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: high risk for ESRD; immunosuppressive treatment; membranous nephropathy; ACTH
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — adrenocorticotropin zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): In this open-label study all patients included are treated in the experimental group.
  Interventions: Drug: tetracosactide hexacetaat

INTERVENTIONS:
Drug: tetracosactide hexacetaat — Intramuscular injections with tetracosactide hexacetaat (Synacthen Depot) 1ml a 1mg/ml. Treatment for 9 months with an increasing dosage from once per 2 weeks to twice a week.
  Other Names: Synacthen Depot, long-acting synthetic ACTH

SUMMARY:
The purpose of this study is to determine whether treatment with long-acting synthetic adrenocorticotropic hormone is in the treatment of patients with idiopathic membranous nephropathy and high for renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven idiopathic membranous nephropathy.
* Nephrotic syndrome: proteinuria > 3.5 g/day and serum albumine < 30 g/l
* Normal or mildly impaired renal function (eGFR > 60 ml/min, MDRD formula)
* High risk for renal failure: beta-2-microglobulin excretion > 500 ng/min
* Relative contra-indication for cyclophosphamide treatment:

  * fertility and wish for (future) family expanding
  * high age ( > 60 years)
  * former cyclophosphamide treatment
  * intolerance to cyclophosphamide

Exclusion Criteria:

* Clinical,biochemical or histological signs of any underlying systemic disease
* Any infectious disease (including latent tuberculosis and/or latent amoebiasis)
* Active gastric or duodenal ulcers
* Pregnancy, lactation, inadequate contraceptives
* Clinical signs of renal vein thrombosis
* Asthma and /or any allergic conditions or hypersensitivity reactions
* Allergic reaction to synthetic ACTH in the past

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Attainability of ACTH therapy with intramuscular injections twice a week for a period of 9 months, measured as the percentage of injections that has been received in line with the treatment schedule. | 9 months

SECONDARY OUTCOMES:
Efficacy of treatment with ACTH: number of remissions of proteinuria at the end of treatment | 9 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jack FM Wetzels, M.D.Ph.D., Study Director — Department of Nephrology, Radboud University; Julia M Hofstra, M.D., Principal Investigator — Department of Nephrology, Radboud University
Locations (1):
- Radboud University, Nijmegen, Netherlands

REFERENCES:
- [Derived] van de Logt AE, Beerenhout CH, Brink HS, van de Kerkhof JJ, Wetzels JF, Hofstra JM. Synthetic ACTH in High Risk Patients with Idiopathic Membranous Nephropathy: A Prospective, Open Label Cohort Study. PLoS One. 2015 Nov 12;10(11):e0142033. doi: 10.1371/journal.pone.0142033. eCollection 2015. PMID 26562836